CLINICAL TRIAL: NCT04794010
Title: A German, Nationwide, Prospective, Observational, Multicenter Study in Patients With First-line Nivolumab Plus Ipilimumab Therapy Combined With Two Cycles of Chemotherapy for Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study in Participants With First-Line Nivolumab Plus Ipilimumb Therapy Combined With Two Cycles of Chemotherapy for Metastatic Non-Small Cell Lung Cancer
Acronym: FINN
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7MA
Record Dates: First submitted 2021-03-10; First posted 2021-03-11 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; NSCLC; Nivolumab; Ipilimumab; Chemotherapy; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with Metastatic Non-Small Cell Lung Cancer

SUMMARY:
The purpose of the study is to collect real-life data during the early post-market authorization approval period in Germany.

The study aims at describing the outcomes, patient characteristics, safety profile, treatment patterns and patient-reported Quality of Life of first-line treatment with nivolumab plus ipilimumab in combination with two cycles of chemo therapy in participants with confirmed stage IV Non-Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV Non-Small Cell Lung Cancer (NSCLC) (histologically or cytologically confirmed stage), without known Epidermal Growth Factor Receptor (EGFR)- or Anaplastic Lymphoma Kinase (ALK)-alterations (according to label approved by EU)
* Decision to initiate a first-line treatment with nivolumab plus ipilimumab combined with two cycles of chemotherapy for the treatment of NSCLC according to the German label has been made independently of the study

Exclusion Criteria:

* Current primary diagnosis of a cancer other than NSCLC that requires systemic or other treatment
* Participants with known EGFR- or ALK-alterations

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is planned to include 825 patients at 100 sites in Germany in this observational study from marketing authorization by the European Medicines Agency (EMA) onwards.
  The planned recruitment phase is approximately 24 months, the planned follow-up phase 60 months from the day of nivolumab plus ipilimumab plus two cycles of chemotherapy initiation (D0).
Sampling Method: Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2027-12-22 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) according to subgroups of interest | Up to 5 years
Progression-free survival (PFS) | Up to 5 years
Duration of treatment | Up to 5 years
Distribution of socio-demographic characteristics of participants | At Baseline
  Age, Sex, Ethnicity, Height, Weight and BMI
Distribution of clinical characteristics of participants | At Baseline
  Histology subtype, Tumor stage, Location or primary tumor and Location of metastases
Description of participant-reported outcomes (PROs) of participants using European Quality of Life-5 Dimensions (EQ-5D) questionnaires | Up to 5 years
Description of participant-reported outcomes (PROs) of participants using Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) | Up to 5 years
Management of AEs: Treatment of AEs | Up to 5 years
Management of AEs: Date of occurrence of AE | Up to 5 years
Management of AEs: Start of treatment | Up to 5 years
Treatment Patterns: Previous therapies | Up to 5 years
Treatment Patterns: Subsequent therapies | Up to 5 years
Treatment patterns: Concomitant medication | Up to 5 years
Treatment patterns : Management of treatment-related adverse events [AEs], previous and subsequent therapies | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Leipzig, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html